CLINICAL TRIAL: NCT05200910
Title: Nutritional, Hormonal and Anthropometric Evaluation of Children After Transcatheter VSD Closure
Brief Title: The Effect of Transcatheter VSD Closure on Children's Appetite, Hormones and Growth
Status: Completed | Type: Observational
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, süleyman sunkak, Specialist (pediatric cardiolog), Kayseri City Hospital
Other Study IDs: 7645
Record Dates: First submitted 2021-12-03; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Ventricular Septal Defect; Appetite Loss; Growth Delay
Keywords: ventricular septal defect; appetite; growth; interventional therapy
MeSH Terms: conditions — Heart Septal Defects, Ventricular; Anorexia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples, plasma, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Patients whose ventricular septal defect closed percutaneously.
- Control: Healthy children

SUMMARY:
In this study; Changes in appetite, hormones and growth of ventricular septal defect patients treated with non-surgical method were evaluated.

DETAILED DESCRIPTION:
The study included 20 patients whose ventricular septal defect closed percutaneously and 26 children as control group. The symptoms, anthropometric measurements and laboratory tests of patient group were recorded at initial, 1st month and 6th months after closure.

Anthropometric measurements; weight for age (WFA), height for age (HFA), body mass index (BMI) and their z scores, triceps skinfold thickness (TSF) and mid-upper arm circumference (MUAC) were recorded on admission. Patients with weight for height z score less than -2 were defined as malnutrition.

Questions about the symptoms like appetite, weight gain, frequency of illness, rate of breathing, fatigue were asked to all parents at initial. These questionnaires15 and visual analogue scale (for appetite) were repeated at 1st and 6th month visits.

During the initial evaluation, approximately 6 ml of venous blood samples were taken between 9:00-10:00 am after an average of 10 hours fasting. On the same day, IGFBP-3, Ghrelin and leptin,fasting blood glucose, insulin, IGF-1, IGFBP-3, aspartate aminotransferase (AST) and alanine aminotransferase (ALT), total protein, and albumin were measured.

Anthropometric measurements and laboratory tests were repeated at 1st and 6th month visits.

ELIGIBILITY:
Inclusion Criteria:

Pediatric patients who underwent transcatheter VSD closure

Exclusion Criteria:

* Chromosomal abnormalities
* Additional systemic disease
* Systemic infections

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric patients who underwent transcatheter VSD closure in our institute and whose growth was followed for 6 months as patient group.
  Healthy children without appetite or growth retardation were included in the study as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Weight Z score | 6 months
  The change in the Z scores of the heights according to the age of the patients after the interventional closure of the VSD
Height Z score | 6 month
  The change in the Z scores of the heights according to the age of the patients after the interventional closure of the VSD
Body mass index Z score | 6 month
  The change in the Z scores of the body mass index according to the age of the patients after the interventional closure of the VSD
Ghrelin | 6 month
  Change in serum ghrelin level of patients after interventional closure of VSD
Leptin | 6 month
  Change in serum leptin level of patients after interventional closure of VSD
Visual analogue scale | 6 month
  Change in Visual analogue scale of patients and parent after interventional closure of VSD. Values in this scale vary between 0-100 mm, values close to '0' are composed of words and images expressing a decrease in the patient's appetite, values close to '100' representing an increase in appetite.

CONTACTS AND LOCATIONS:
Overall Officials: Onur Tasci, Principal Investigator — TC Erciyes University
Locations (1):
- Süleyman Sunkak, Kayseri, Kocasinan, Turkey (Türkiye)